CLINICAL TRIAL: NCT05694273
Title: Acute Cerebrovascular Events in Patients Undergoing Catheter Ablation (CENTRAL): an Investigator-initiated, Multicenter Real-world Study
Brief Title: Acute Cerebrovascular Events in Patients Undergoing Catheter Ablation
Acronym: CENTRAL
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Shaanxi Provincial People's Hospital (Other); 521 Hospital of NORINCO Group (Other); Xiangyang Central Hospital (Other); Ankang Central Hospital (Other); Baoji Central Hospital (Other); Luoyang Central Hospital (Other); Tianjin Medical University Second Hospital (Other); Fu Wai Hospital, Beijing, China (Other); Fuwai Yunnan Cardiovascular Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-531
Record Dates: First submitted 2023-01-10; First posted 2023-01-23 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Arrhythmia; Acute Cerebrovascular Disease
Keywords: Catheter ablation; Arrhythmia; Major adverse cardiovascular and cerebrovascular events (MACCE)
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ischemic stroke group: 1. Ischemic stroke secondary to patients receiving catheter ablation.
  2. Ischemic stroke met the diagnostic criteria of the 2018 edition of the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke, and was confirmed by cranial CT/MRI scan.
- Transient ischemic attack group: 1. Transient ischemic attack secondary to patients receiving catheter ablation.
  2. Ischemic stroke met the diagnostic criteria of the 2018 edition of the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke, and was confirmed negative of new onset of infarction by cranial CT/MRI scan.
- Cerebral hemorrhage group: 1. Cerebral hemorrhage secondary to patients receiving catheter ablation.
  2. Cerebral hemorrhage met the diagnostic criteria of the 2021 Chinese Guidelines for the Diagnosis and Treatment of cerebral hemorrhage and was confirmed by head CT/MRI.
- Contral group: Patients who did not experience acute cerebrovascular events in the hospital.

SUMMARY:
This study aims to evaluate the incidence, clinical characteristics, and short-term prognosis of acute cerebrovascular events occurring in-hospital in patients with arrhythmias following catheter ablation. The goal is to provide evidence supporting the improvement of patient quality of life and reduction of in-hospital acute cerebrovascular complications in patients with post-ablation arrhythmias. This will also contribute to the evidence-based clinical management of such patients.

DETAILED DESCRIPTION:
With the steady development of catheter ablation, it has gradually become the main treatment of various arrhythmias. Antithrombotic and anticoagulant therapy after catheter ablation determines the occurrence of perioperative bleeding and ischemic events. However, the incidence, characteristics and short-term prognosis of secondary acute cerebrovascular events in patients with arrhythmia after catheter ablation have not been studied. Methods: This study was intended to retrospectively collect and analyze the case data and auxiliary examination results of patients with arrhythmia who underwent catheter ablation. To evaluate the incidence, clinical features and short-term prognosis of secondary acute ischemic and hemorrhagic cerebrovascular events in patients with arrhythmia after catheter ablation. In order to improve the quality of life of patients, reduce the secondary acute cerebrovascular complications in the hospital in patients with arrhythmia after catheter ablation, to provide evidence for promoting the clinical management of such patients, and to provide help for the maximum degree of prevention and control risk.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients who undergo catheter ablation for arrhythmias.

Exclusion Criteria:

* 1. Patients were diagnosed of acute cerebrovascular disease prior to radiofrequency catheter ablation;
* 2. Patients < 18 years or > 80 years;
* 3. Patients with uncomplete clinical data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plans to enroll patients with arrhythmias who undergo catheter ablation and meet the specified inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of MACCE | 3 months after enrollment
  Major adverse cardiovascular and cerebrovascular events, a composite of all-cause mortality, myocardial infarction and stroke. The data will be obtained at 3-month follow-up, according to medical records of all patients.

SECONDARY OUTCOMES:
Incidence of all-cause mortality | 3 months after enrollment
  The data will be obtained at 3-month follow-up, according to medical records of all patients.
Incidence of myocardial infarction | 3 months after enrollment
  The data will be obtained at 3-month follow-up, according to medical records of all patients.
Incidence of stroke | 3 months after enrollment
  The data will be obtained at 3-month follow-up, according to medical records of all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided